CLINICAL TRIAL: NCT06421337
Title: Somatosensory Evoked Potential (SEP) N20 Monitoring With BraiN20® Medical Device for Prediction of Functional Independence Defined as Rankin Scale Score 0-2 in Global Patients With Suspected Acute Stroke.
Brief Title: BraiN20® Medical Device in Suspected Acute Stroke Patients
Acronym: PROMISE-GLOB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alicia Martínez Piñeiro (Other)
Responsible Party: Sponsor-Investigator, Alicia Martínez Piñeiro, Principal Investigator, Fundació Institut Germans Trias i Pujol
Organization: Fundació Institut Germans Trias i Pujol (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROMISE GLOBAL CIP V2.0
Record Dates: First submitted 2024-04-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Acute Stroke
Keywords: Somatosensory evoked potentials; Acute stroke ischemic; Acute stroke hemorrhagic; Stroke mimics; Prognosis; Functional recovery; Medical device; Diagnostic
MeSH Terms: conditions — Stroke; Ischemic Stroke; Disease

STUDY DESIGN:
Masking Description: Outcome will be evaluated by an independent assessor blinded to the monitoring results at the acute phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Subjects presenting at emergency departments of participating hospitals with suspected acute stroke within 24 hours from symptom onset with or without stroke code activation
  Interventions: Device: BraiN20(R)

INTERVENTIONS:
Device: BraiN20(R) — SEP monitoring will be carried out using the BraiN20® medical device and appropriate electrodes. SEP of both median nerves will be recorded, transferred, and stored to the internal card for their evaluation. BraiN20® Medical Device provides an automatic reading of the presence and feature of a N20 response both ipsilateral and contralateral (as control) to the cerebral hemisphere affected by the stroke and do not require specific training. Furthermore, the device provides an outcome prediction (percentage of likelihood of having mRS ≤ 2 day 7 and 90 after stroke onset) based on an internal algorithm.
  BraiN20® measures one N20 wave per 33 seconds. Scalp electrodes are easily embedded on a headband and the wrist electrodes on a glove.

SUMMARY:
Time is Brain company (http://www.tibtimeisbrain.com/about_us/) developed BraiN20®, a medical device to assess the presence and characteristics of the N20 signal of SEP. Investigators have demonstrated a high prognostic accuracy of N20 on functional recovery of patients with acute ischemic stroke (AIS) due to large vessel occlusion (LVO) undergoing endovascular thrombectomy (EVT), the gold standard treatment. The aim if this new project is to validate BraiN20® in global patients presenting with suspected acute ischemic or hemorrhagic stroke in three comprehensive stroke centers in Spain. The primary objective is to establish the predictive performance of the presence of the N20 SEP over functional recovery as the primary outcome measure (likelihood of having a modified Rankin Scale (mRS) score 0-2 at 3 months evaluated by blinded independent raters). The effect will be measured by the metrics sensitivity, specificity, and predictive values, and compared with clinical and imaging predictive models by Receiving Operating Characteristics (ROC) curve analysis in the global population, stroke subtype and stroke mimics. Secondary aims are: 1) to determine the area under the curve (AUC) of the presence of the N20 SEP as biomarker of functional recovery in small subcortical infarctions and in patients with cortical infarctions and no large vessel occlusion; 2) to characterize N20 SEP signal in hemorrhagic stroke and stroke mimics; and 3) to evaluate the discriminant capacity of an explanatory new algorithm combining pre-hospital clinical variables and N20-SEP signal characteristics between ischemic, hemorrhagic and stroke mimics.

This project would represent the first pilot study to validate the ability of BraiN20® to predict the functional recovery in the different types of acute stroke but also its ability to discriminate between stroke subtypes. Thus, BraiN20® monitoring could arise as a paradigm shift in acute stroke management, since it would standardize and accelerate patient triage, enable real time monitoring, increase access to EVT treatment and improve its outcome The trial is sponsored by Time is Brain S.L. and started in March 2024. Primary endpoint results are expected by the end of the 2024.

BraiN20® could be a useful medical device aiding stroke subtype diagnosis and functional recovery.

DETAILED DESCRIPTION:
The likelihood of a favourable outcome of acute stroke is critically dependent on patients presenting promptly after symptom onset and on hospitals providing immediate access to the gold standard treatment: the EVT. The current clinical stroke management is complex, time-consuming, requires different hospital settings with specialized equipment, and diagnostic is based on momentaneous snapshot providing brain imaging and clinical scores, without real-time monitoring tools. In addition, the current standard of care is unfavourable to patients localized far from a Comprehensive Stroke Center (CSC), especially for those living in rural regions. Thus, 50% undergoing EVT do not respond to the treatment because their brain tissue has been already irreversibly damaged.

Thus, neurologists from the Germans Trias I Pujol CSC (Barcelona, Spain) started a new research line by introducing a new diagnostic approach based on neurophysiological techniques to optimize the selection of patients benefiting from EVT and improve its outcome. In 2018, the Somatosensory Evoked Potentials MonItoring During Acute Ischemic Stroke (PROMISE) clinical trial confirmed in a large cohort (n=228) that the N20 SEP determined before EVT increases 30% the diagnostic accuracy of salvageable brain compared to the technologies currently used.

Time is Brain S.L. (TiB) was founded in July 2020 by neurologists from Germans Trias I Pujol CSC to develop BraiN20®, a medical device to assess presence and characteristics of N20 SEP signal from AIS onset and during the entire stroke patient journey. It promises to be an accurate, relatively inexpensive, userfriendly device to quickly determine N20 signal of the SEPs. This technology is safe and non-invasive and therefore may be especially useful at the pre-hospital stage of stroke patients, monitoring brain viability in-hospital and in particular in the angio-room guiding therapeutic strategies.

PROMISE20 (Somatosensory Evoked Potentials Monitoring in Patients with Acute Ischemic Stroke and Large Anterior Vessel Occlusion Undergoing Endovascular Thrombectomy. A Clinical Validation of the BraiN20® Medical Device) (NCT06149754) is underway.

The primary aim is to prove that the percentage of patients with optimal or good reliability of the BraiN20® Medical Device automatic recording of N20 is higher than 75% (i.e., the lower limit of the one-sided 95% confidence interval is higher or equal to 75%), assuming a true proportion equal to 87.5%, according to the classification by two expert physicians blind to BraiN20® reading results.

While the usefulness of N20 SEP in AIS patients undergoing EVT has already been demonstrated, the predictive performance of BraiN20® is unknown in other stroke subtypes and stroke mimics. This project aims to validate for the first time BraiN20® monitoring in global patients presenting with suspected acute ischemic or hemorrhagic stroke. The accomplishments so far make a strongly believe that BraiN20® will enable a step improvement and become the cornerstone of the acute stroke patient journey

The study will investigate the ability of the BraiN20® medical device to detect and characterize N20 signal in a global population of suspected stroke patients.

The primary objective is to establish the predictive performance of the presence of N20 SEP registered by BraiN20® over functional recovery (primary outcome) (likelihood of having a mRS score 0-2 at 90 days evaluated by blinded independent raters). The effect will be measure by the metrics sensitivity, specificity and predictive values, and compared with clinical and imaging predictive models by ROC curve analysis in the global population, stroke subtypes and stroke mimics.

Secondary aims are:

* to determine the area under the AUC of the N20 amplitude predicting functional recovery in small subcortical infarctions and in patients with spontaneous LVO revascularization.
* to characterize N20 signal in intracranial hemorrhage (ICH) and stroke mimics.
* to evaluate the discriminant capacity of an explanatory new algorithm combining prehospital clinical variables and N20 signal characteristics between ischemic stroke, ICH and stroke mimics.
* to characterize N20 signal in posterior ischemic strokes and basilar occlusion.

Safety outcomes related to BraiN20® monitoring are:

* Frequency of patients in whom N20+ recording prior to treatment disappears after specific treatment such as thrombectomy procedure, or surgical treatment.
* Mortality at day 7.
* Tolerability of the BraiN20® monitoring.
* Number of consumables used with mean and standard deviation

PROMISE-GLOB is a prospective, interventional, single arm, multi-center, open trial with blinded evaluation of the primary endpoint of a cohort of patients with suspected acute stroke admitted in the emergency department of a CSC. The study will be performed in consecutive patients fulfilling eligibility criteria in three comprehensive stroke centers in Spain.

Patients will be studied and managed according to local protocols. No special recommendations are given, but protocols must define criteria for acute medical treatment, intravenous thrombolysis, endovascular thrombectomy, hemicraniectomy and surgical evacuation of ICH. Regarding diagnostic tools, computed tomography (CT), CT angiography (CTA), magnetic resonance (MR) or MR angiography (MRA) and ultrasound will be used at discretion of investigators for a required classification of stroke subtype or stroke mimics.

SEP monitoring with the BraiN20® medical device will be performed as soon as possible after admission preferably before IV thrombolysis as long as it does not entail a delay in the acute emergency therapies. In patients undergoing EVT or surgical therapies, baseline SEP monitoring should be performed before these procedures, and repeated at the end of them. SEP monitoring should also be repeated in case of neurologic deterioration ≥ 4 points in the National Institute of Health Stroke Scale (NIHSS) within the first 24 hours.

Patients' cohort will be followed up to 90 days after inclusion. mRS score will be determined at day 7 or discharge and at day 90 by a local investigator blind to the BraiN20® recordings, both face to face or by telephone interview. There are no specific study interventions. Patients will be discharged at home, other centers or admitted at acute stroke units (or intensive care units if needed) and treated following the European Stroke Organization guidelines.

SEP monitoring will be carried out using the BraiN20® medical device and appropriate electrodes. SEP of both median nerves will be recorded, transferred, and stored to the internal card for their evaluation. BraiN20® Medical Device provides an automatic reading of the presence and feature of a N20 response both ipsilateral and contralateral (as control) to the cerebral hemisphere affected by the stroke and do not require specific training. Furthermore, the device provides an outcome prediction (percentage of likelihood of having mRS ≤ 2 day 7 and 90 after stroke onset) based on an internal algorithm. BraiN20® measures one N20 wave per 33 seconds. Scalp electrodes are easily embedded on a headband and the wrist electrodes on a glove.

SEP recording will be done in the emergency room or in the angiography or surgical room (if required). Examiners will be physicians or nurses in charge of the patient. N20 recordings will be stored in the device for review at the end of the trial. It is recommended to obtain three recordings of the N20 response to confirm its presence or absence and exclude a noisy registration in the affected side (this takes approximately 3 min). Presence of the N20 response in the contralateral side will be used as control to rule out technical issues or the effect of other conditions that could affect the SEPs recordings.

At admission at the Emergency Unit, patients with suspected acute stroke will be immediately attended by neurologists. NIHSS will be evaluated, blood will be drawn for baseline analysis and CT/CTA neuroimaging performed if indicated by local protocols. Anytime during these procedures BraiN20® electrodes will be placed and three N20 recordings obtained from each brain side (stroke side and control hemisphere). Serum glucose, body temperature and blood pressure will be controlled following the American Stroke Association guidelines. Alberta Stroke Program Early CT (ASPECT) score, ICH volume (AxBxC/2) and location will be measured by local investigators on baseline CT. Informed consent either, oral, signed or deferred will be obtained.

Stroke subtype will be classified according to the Oxfordshire Community Stroke Project (OCSP) complemented with neuroimaging findings as total anterior cerebral infarction (TACI), partial anterior cerebral infarction (PACI), posterior cerebral infarction (POCI) and lacunar infarction (LACI); in addition deep ICH and lobar ICH. Stroke etiology following the classification of the Cerebrovascular Diseases Study Group of the Spanish Neurological Society as small vessel disease, large artery atherosclerosis (extracranial or intracranial), atrial fibrillation (AF) or other cardioembolic diseases, Unknown, Other (e.i. arterial dissection) and stroke mimic.

A specific case record form (CRF) will be generated for each eligible patient. The completion of the CRF will be made by authorized site personnel. A copy of the CRF will be kept in the hospital records and the original will be collected by the sponsor. The investigator must ensure the accuracy, completeness and timeliness of data reported in the CRF. The sponsor will test all data for completeness, consistency, and plausibility, and produce queries for erroneous, incomplete and missing data. Any necessary queries will be sent to the investigator by email. Periodic monitoring visits will be made by the sponsor throughout the investigation to ensure that the investigator's obligations are being fulfilled. The database will be keep anonymized and confidentially at the sponsor workplace for centralized monitoring of the electronic records. Resolved queries will be returned to the sponsor by email. If answers are incomplete or discrepant with other data, re-queries may be necessary.

No a priori sample size calculation has been done because it is unknown the potential predictive capacity of BraiN20® in a non-selected stroke population. This population has not been previously studied and this pilot study aims to establish the proof of concept for a future phase III design. The study period is limited to 8-12 months inclusion in three stroke centers and 500 evaluable patients are expected. This sample size is appropriate for including more than 100 patients in each stroke subtype. Patients that do not fulfil eligibility criteria will be replaced in order to obtain 500 evaluable patients.

No risk or benefit for patients is expected in the trial since it is an study without any specific decision-making based on the BraiN20® results. Any device malfunction or unexpected characteristics will be registered, and the device unit discarded (returned to Time is Brain, S.L. for inspection).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected acute stroke ischemic or hemorrhagic admitted in the emergency department within 24 hours from symptoms onset or from the last time seen normal.
2. Stroke mimics classified after neurologic examination and diagnostic procedures will be also included.
3. Age ≥18.
4. No significant pre-stroke functional dependence (mRS ≤ 2).
5. Baseline NIHSS score obtained prior to procedure must be equal or higher than 1 point. Patients with TIA and full recovery on admission must not be included.
6. Patients in whom BraiN20® monitoring can be performed without delay of acute stroke therapies.
7. Participation in other treatment or diagnostic test clinical trial is allowed if the patients fulfill the inclusion criteria of PROMISE-GLOBAL.
8. Informed consent obtained from patient or acceptable patient surrogate; or the deferred informed consent, to avoid the delay in the start of the stroke emergency therapies.

Exclusion Criteria:

- Clinical criteria

1. Patients with a well-documented history of neuromuscular diseases and other severe neurodegenerative disorders (Mild Cognitive Impairment is not exclusion criteria), prior stroke (TIA is not exclusion criteria) or nervous system tumors that could interfere with SEP assessment.
2. Serious, advanced, or terminal illness with an anticipated life expectancy of less than three months.
3. Women in the premenopausal period.

   - Neuroimaging criteria
4. Acute infarct volume (ASPECTS) or ICH volume (AxBxC/2) on plane CT should be measured but they are not exclusion criteria and should not preclude any specific treatment according to local protocols (i.e., mechanical thrombectomy, hemicraniectomy or ICH evacuation).
5. Evidence of intracranial tumor (except small meningioma).

   - BraiN20® medical device safety issues:
6. Subjects with a demand-type cardiac pacemaker, defibrillator, or other electrical implant or metal.
7. Patients with suspected or well-known cancerous skin lesions in the area where electrical stimulation is to be applied.
8. Patients who have a localized disorder in the wrist and forearm where electrical stimulation is to be applied (i.e., fractures or dislocations, vein puncture).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Functional recovery at 3 months | Day 90
  Functional recovery is defined by modified Rankin Scale score 0-2 (min 0, no disability; max 6, death) at day 90 after stroke. Modified Rankin Scale score will be measured by blinded local raters according to a structured interview at day 7 or before discharge and at day 90 by telephone interview or face to face. Two cohort groups are defined:
  Stroke functional recovery: mRS lower or equal than 2 at 90 ± 15 days. Stroke functional dependence: mRS higher than 2 at 90 ± 15 days.

SECONDARY OUTCOMES:
N20 signal characteristics | At admission within 24 hours from stroke onset
  Amplitude, latency and wave characteristics of the N20 response will be used to make a new algorithm able to discriminate between ischemic, hemorrhagic and stroke mimics.
National Institute of Health Stroke Scale score (NIHSS) | Days 7 and 90
  Evaluation of the severity of the focal neurologic deficit (NIHSS: min 0, no neurological deficit; max 42)

OTHER OUTCOMES:
Tolerability of the BraiN20® monitoring | At admission within 24 hours from stroke onset
  Comfortability of the patients during the 3-5 minutes of monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Dávalos, MD, PhD, Study Chair — Fundació Institut d'Investigació en Ciències de la Salut Germans Trias iPujol
Locations (3):
- Spain (3):
  - Hospital Universitari de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: No
Result will be presented at the European Stroke Organization Conference and published

REFERENCES:
- [Background] Alicia Martinez-Piñeiro MD, PhD aliciamp@tibtimeisbrain.com , Giuseppe Lucente MD, PhD , María Hernandez-Perez MD, PhD , Jordi Cortés PhD , Andrea Arbex MD , Natalia Pérez de la Ossa MD, PhD , Alba Ramos-Fransí MD, PhD , Miriam Almendrote MD , Mònica Millán MD, PhD , Meritxell Gomis MD, PhD , Laura Dorado MD, PhD , Carlos Castaño MD, PhD , Sebastián Remollo MD , Patricia Cuadras MD, PhD , Alicia Garrido MD , Nicolau Guanyabens MD , Joaquim Broto MD , Elena López-Cancio MD, PhD , Jaume Coll-Canti MD, PhD , Antoni Dávalos MD, PhD , and PROMISE (Somatosensory Evoked POtEntials MonItoring During Acute Ischemic StrokE) Study Group. Prognostic Accuracy of N20 Somatosensory Potential in Patients With Acute Ischemic Stroke and Endovascular Thrombectomy. Stroke: Vascular and Interventional Neurology. 2023 | Volume 3, Issue 5: e000735
- [Background] Pittock SJ, Meldrum D, Hardiman O, Thornton J, Brennan P, Moroney JT. The Oxfordshire Community Stroke Project classification: correlation with imaging, associated complications, and prediction of outcome in acute ischemic stroke. J Stroke Cerebrovasc Dis. 2003 Jan;12(1):1-7. doi: 10.1053/jscd.2003.7. PMID 17903897
- [Background] Sobrino Garcia P, Garcia Pastor A, Garcia Arratibel A, Vicente Peracho G, Rodriguez Cruz PM, Perez Sanchez JR, Diaz Otero F, Vazquez Alen P, Villanueva Osorio JA, Gil Nunez A. [Aetiological classification of ischaemic strokes: comparison of the new A-S-C-O classification and the classification by the Spanish Society of Neurology's Cerebrovascular Disease Study Group]. Neurologia. 2013 Sep;28(7):417-24. doi: 10.1016/j.nrl.2012.07.005. Epub 2012 Sep 19. Spanish. PMID 22998938
- See also: Startup developing BraiN20(R) — http://timeisbrain.com